CLINICAL TRIAL: NCT02644109
Title: Effect On Serum Cholesterol Of Dairy Products With Addition Of Esterified Phytosterols In Chilean Subjects With Hypercholesterolemia
Brief Title: Effect On Serum Cholesterol Of Dairy Products With Addition Of Esterified Phytosterols
Acronym: ACTICOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Natalia Jara, MD, MSc, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Acticol - 001
Record Dates: First submitted 2015-12-21; First posted 2015-12-31 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-08

CONDITIONS: Dyslipidemias; Hypercholesterolemia
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia | interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phytosterols (Experimental): 1. Milk powder: subjects will be instructed to consume 22 g/day of the product, with 0.65 g of esterified phytosterols (0.39 g of free equivalent sterols). The product will be reconstituted with 200 ml of water at time of consumption, preferably at breakfast or tea time. The total amount of product will be provided at the beginning of the study (day 1), together with instructions, material for preparation, and storage.
  2. Drinking yoghurt: the daily volume consumed will be 90 ml/day with 1.3 grs of esterified phytosterols (0.78 g of free equivalent phytosterols). Subjects will be instructed to consume this beverage with main meal (not later than 15 min after it. The product should be kept refrigerated. Products will be distributed to subjects on a weekly basis.
  Interventions: Dietary Supplement: Phytosterol
- Placebo (Placebo Comparator): 1. Milk powder: subjects will be instructed to consume 22 g/day of the product, without phytosterols. The product will be reconstituted with 200 ml of water at time of consumption, preferably at breakfast or tea time. The total amount of product will be provided at the beginning of the study (day 1), together with instructions, material for preparation, and storage.
  2. Drinking yoghurt: the daily volume consumed will be 90 ml/day without phytosterols. Subjects will be instructed to consume this beverage with main meal (not later than 15 min after it. The product should be kept refrigerated. Products will be distributed to subjects on a weekly basis.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Phytosterol — Day 1: Anthropometry, laboratory test, dietary intake (24 hour recall and food frequency questionnaire) and presence of symptoms and side effects will be determined, a logbook will be provided to record product consumption, symptoms, medications and side effects. Then will be randomly assigned to one of the groups.
  Days 7 & 21: 24 hour recall, review of symptoms, side effects and adherence as registered in the logbook.
  Days 15 & 30: Anthropometry, vital signs, venous blood sample, review of symptoms, side effects and adherence to intervention as registered on logbook, dietary intake (24-hour recall), delivery of monetary compensation proportional to the study days will be given before being discharged.
  Other Names: ACTICOL
  Arms: Phytosterols
Dietary Supplement: Placebo — Day 1: Anthropometry, laboratory test, dietary intake (24 hour recall and food frequency questionnaire) and presence of symptoms and side effects will be determined, a logbook will be provided to record product consumption, symptoms, medications and side effects. Then will be randomly assigned to one of the groups.
  Days 7 & 21: 24 hour recall, review of symptoms, side effects and adherence as registered in the logbook.
  Days 15 & 30: Anthropometry, vital signs, venous blood sample, review of symptoms, side effects and adherence to intervention as registered on logbook, dietary intake (24-hour recall), delivery of monetary compensation proportional to the study days will be given before being discharged.
  Arms: Placebo

SUMMARY:
Hypercholesterolemia is an important risk factor for cardiovascular disease, asociated primarily with high plasma levels of LDL lipoprotein, which in turn depend on the endogenous hepatic synthesis of cholesterol and its absorption at intestinal level. It has been demonstrated that there reducing plasma LDL is beneficial, mainly with the use of statins, which are the first treatment option for a moderate hypercholesterolemia.

Phytosterols reduce the intestinal absorption of cholesterol by reducing its incorporation into lipid micelles. Consequently, phytosterols have become a relevant alternative treatment against low hypercholesterolemia. The target population are 40 to 65 years old individuals with low hypercholesterolemia.

DETAILED DESCRIPTION:
Different protocols have demonstrated that phytosterol intake fluctuates between 1000 to 2000 mg per day decreasing LDL by around 10%, independently of levels of blood triglycerides and HDL (high density lipoproteins) concentrations. In fact, the National Cholesterol Education Program and the American Heart Association recommend the addition of 2 g/day of phytosterols to daily diet of adults. This is also recommended by the FDA (Food and Drug administration).

Phytosterols delivery has been proven effective when administrated in lipid matrixes such as margarines and dressings and low-fat such as skimmed milk and yogurt, proving to have an hypolipidemic effect. The investigational products consist of powder milk and a drinking yoghurt with the addition of esterified phytosterols, with a total daily intake of 1.95 g/day (1.17 g/day of free equivalent).

Primary objective: To evaluate the impact in Chilean population of phytosterols incorporated into dairy products in reduction of LDL cholesterol.

Secondary objectives:

1. To evaluate potential changes in blood cholesterol concentration according to nutritional state and age.
2. To determine the appearance of symptoms and/or effects during the intervention period.

The trial has been designed to evaluate the effect of phytosterols incorporated to low fat dairy products in Chile, through the consumption of one glass of milk powder and 90 mL of drinking yoghurt, which results in a daily consumption of 1.95 g/day of esterified phytosterols. This amount falls within demonstrated effective doses reported in literature.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between 40 to 65 y old.
2. Males and females.
3. Body mass index between 20 to 35 kg/m2
4. Mild hypercholesterolemia (LDL between 130 to 190 mg/dl) without requirement of immediate pharmacological treatment.
5. Without symptoms of atherosclerotic vascular disease.
6. Regular consumption of dairy foods (at least once a day).
7. Sedentary lifestyle defined as less than 20 min, three times per week of moderate to intense physical activity)

Exclusion Criteria:

1. Individuals with sitosterolemia.
2. Use of hypolipidemic drugs within the past 6 weeks before initiated the study.
3. Presence of type 1 or 2 diabetes; nephrotic syndrome or chronic kidney disease at stage III (estimated glomerular filtration rate<60 ml/min) or higher; gastrointestinal, liver, hepatobiliary, endocrine diseases or any condition potentially effecting lipid metabolism.
4. History of heart failure, unstable angina, cerebrovascular accident, heart failure, uncontrolled arrhythmias, high blood pressure (systolic>160 mm/Hg or diastolic>100 mm/Hg), cardiac surgery or other vascularization procedure.
5. Blood triglycerides higher than 400 mg/dl.
6. History of cancer disease over the last 5 years.
7. Pregnant and lactating women.
8. Lactose intolerant individuals or presence of related symptoms
9. Individuals with cow´s milk protein allergy.
10. Vegetarians
11. Regular use of drugs for obesity treatment, or affecting lipid metabolism.
12. Regular use of nutritional supplements.
13. Smokers having more than 5 units per day.
14. Individuals drinking more than 3 standard units per day of alcoholic beverages (>3 glasses of wine, 2 beers o 1 strong alcohol).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Hirsch, MD, Study Director — University of Chile
Locations (2):
- Chile (2):
  - Department of Nutrition, Diabetes and Metabolism. Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan
  - Instituto de Nutricion y Tecnologia de los Alimentos, Universidad de Chile, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Goff DC Jr, Lloyd-Jones DM, Smith SC Jr, Blum C, Schwartz JS; 2013 ACC/AHA Cholesterol Guideline Panel. Treatment of blood cholesterol to reduce atherosclerotic cardiovascular disease risk in adults: synopsis of the 2013 American College of Cardiology/American Heart Association cholesterol guideline. Ann Intern Med. 2014 Mar 4;160(5):339-43. doi: 10.7326/M14-0126. PMID 24474185
- [Result] Korpela R, Tuomilehto J, Hogstrom P, Seppo L, Piironen V, Salo-Vaananen P, Toivo J, Lamberg-Allardt C, Karkkainen M, Outila T, Sundvall J, Vilkkila S, Tikkanen MJ. Safety aspects and cholesterol-lowering efficacy of low fat dairy products containing plant sterols. Eur J Clin Nutr. 2006 May;60(5):633-42. doi: 10.1038/sj.ejcn.1602362. PMID 16404415
- [Result] Mannarino E, Pirro M, Cortese C, Lupattelli G, Siepi D, Mezzetti A, Bertolini S, Parillo M, Fellin R, Pujia A, Averna M, Nicolle C, Notarbartolo A. Effects of a phytosterol-enriched dairy product on lipids, sterols and 8-isoprostane in hypercholesterolemic patients: a multicenter Italian study. Nutr Metab Cardiovasc Dis. 2009 Feb;19(2):84-90. doi: 10.1016/j.numecd.2008.03.012. Epub 2008 Aug 31. PMID 18762410
- [Result] Ortega RM, Palencia A, Lopez-Sobaler AM. Improvement of cholesterol levels and reduction of cardiovascular risk via the consumption of phytosterols. Br J Nutr. 2006 Aug;96 Suppl 1:S89-93. doi: 10.1079/bjn20061708. PMID 16923260
- [Result] Nestel P, Cehun M, Pomeroy S, Abbey M, Weldon G. Cholesterol-lowering effects of plant sterol esters and non-esterified stanols in margarine, butter and low-fat foods. Eur J Clin Nutr. 2001 Dec;55(12):1084-90. doi: 10.1038/sj.ejcn.1601264. PMID 11781675
- [Result] Miettinen TA, Puska P, Gylling H, Vanhanen H, Vartiainen E. Reduction of serum cholesterol with sitostanol-ester margarine in a mildly hypercholesterolemic population. N Engl J Med. 1995 Nov 16;333(20):1308-12. doi: 10.1056/NEJM199511163332002. PMID 7566021

RESULTS

PARTICIPANT FLOW:
Groups:
- Phytosterols: 1. Milk powder: subjects will consume 22 g/day of the product, with 0.65 g of esterified phytosterols (0.39 g of free equivalent sterols). The product will be reconstituted with 200 ml of water at time of consumption.
  2. Drinking yoghurt: the daily volume consumed will be 90 ml/day with 1.3 grs of esterified phytosterols (0.78 g of free equivalent phytosterols).
  Day 1: Anthropometry, laboratory test, dietary intake (24 hour recall and food frequency questionnaire), presence of symptoms and side effects will be determined. Then will be randomly assigned to one of the groups.
  Days 7 & 21: 24 hour recall, review of symptoms, side effects and adherence as registered in the logbook.
  Days 15 & 30: Anthropometry, vital signs, venous blood sample, review of symptoms, side effects and adherence to intervention as registered on logbook, dietary intake (24-hour recall), delivery of monetary compensation proportional to the study days will be given before being discharged.
- Placebo: 1. Milk powder: subjects will be instructed to consume 22 g/day of the product, without phytosterols. The product will be reconstituted with 200 ml of water at time of consumption.
  2. Drinking yoghurt: the daily volume consumed will be 90 ml/day without phytosterols.
  Day 1: Anthropometry, laboratory test, dietary intake (24 hour recall and food frequency questionnaire) and presence of symptoms and side effects will be determined, a logbook will be provided to record product consumption, symptoms, medications and side effects. Then will be randomly assigned to one of the groups.
  Days 7 & 21: 24 hour recall, review of symptoms, side effects and adherence as registered in the logbook.
  Days 15 & 30: Anthropometry, vital signs, venous blood sample, review of symptoms, side effects and adherence to intervention as registered on logbook, dietary intake (24-hour recall), delivery of monetary compensation proportional to the study days will be given before being discharged.
Period: Overall Study
Arm/Group | Phytosterols | Placebo
Started | 24 | 28
Completed | 24 | 24
Not Completed | 0 | 4
Not completed — Adverse Event | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phytosterols | Placebo | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (6.1) | 53.2 (6.6) | 53.2 (6.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 7 | 14 | 21
Region of Enrollment [Number; unit: participants]
  Chile | 24 | 28 | 52
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.9 (3.5) | 27.9 (3.2) | 27.9 (3.3)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 231.9 (22.9) | 226.4 (19.3) | 228.9 (21)
LDL-cholesterol [Mean (Standard Deviation); unit: mg/dl] | 149.5 (18.6) | 146.3 (15.6) | 147.7 (16.9)

OUTCOME MEASURES:

1. Primary Outcome: Serum LDL Cholesterol
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Phytosterols | Placebo
Number analyzed (Participants) | 24 | 24
mg/dl | 122.2 (34.6) | 113.5 (33.8)

ADVERSE EVENTS:
Arm/Group | Phytosterols | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/28
Other Adverse Events (participants affected / at risk) | 0/24 | 2/28
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phytosterols (N=24) | Placebo (N=28)
Abdominal pain and bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
urticarial rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior authorization of the text by the Sponsor